CLINICAL TRIAL: NCT02415595
Title: A Phase 2b Randomized, Active-Controlled, Double-Blind Trial to Investigate Safety, Efficacy, and Dose-response of BMS-955176, Given on a Backbone of Tenofovir/Emtricitabine, in Treatment-Naive HIV-1 Infected Adults
Brief Title: Dose-finding Study of BMS-955176 to Treat HIV-1 Infected Treatment-naive Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial ended early due to GI intolerability and treatment-emergent resistance.
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 205891; 2013-005487-26 (EudraCT Number); AI468-038 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2015-03-11; First posted 2015-04-14 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — BMS-955176

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: BMS-955176 60 mg + TDF/FTC (Experimental): BMS-955176 at 60 mg active dose per day + BMS-955176 placebo matching 120 mg + efavirenz (EFV) placebo matching 600 mg + tenofovir/emtricitabine (TDF/FTC) 300/200 mg per day, orally
  Interventions: Drug: BMS-955176; Drug: TDF/FTC
- Arm 2: BMS-955176 120 mg + TDF/FTC (Experimental): BMS-955176 placebo matching 60 mg + BMS-955176 at 120mg active dose per day + EFV placebo matching 600mg + TDF/FTC 300/200mg per day, orally
  Interventions: Drug: BMS-955176; Drug: TDF/FTC
- Arm 3: BMS-955176 180 mg + TDF/FTC (Experimental): BMS-955176 at 60mg active dose per day + BMS-955176 at 120mg active dose per day + EFV placebo matching 600mg + TDF/FTC at 300/200mg per day, orally
  Interventions: Drug: BMS-955176; Drug: TDF/FTC
- Arm 4: EFV + TDF/FTC (Active Comparator): BMS-955176 placebo matching 60mg + BMS-955176 placebo matching 120mg + EFV at 600mg per day + TDF/FTC 300/200mg per day
  Interventions: Drug: EFV; Drug: TDF/FTC

INTERVENTIONS:
Drug: BMS-955176 — HIV Maturation Inhibitor
  Arms: Arm 1: BMS-955176 60 mg + TDF/FTC; Arm 2: BMS-955176 120 mg + TDF/FTC; Arm 3: BMS-955176 180 mg + TDF/FTC
Drug: EFV — EFV
  Arms: Arm 4: EFV + TDF/FTC
Drug: TDF/FTC — TDF/FTC

SUMMARY:
The purpose of this study is to find at least one dose of BMS-955176 that will be safe, effective and tolerable for HIV-1 infected treatment naive adults.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Men and non-pregnant women, at least 18 years of age
* Antiretroviral treatment-naïve; defined as no current or previous exposure to > 1 week of an antiretroviral drug
* Plasma HIV-1 RNA ≥ 1000 copies/mL
* CD4 T-cell count > 200 cells/mm3

Exclusion Criteria:

* Resistance or partial resistance to any study drug determined by tests at Screening
* Current or historical genotypic and/or phenotypic drug resistance testing showing certain resistance mutations to EFV, TDF, FTC, Protease Inhibitors
* Chronic hepatitis B virus (HBV)/ hepatitis C virus (HCV)
* Blood tests that indicate normal liver function
* Hemoglobin < 8.0 g/dL, platelets < 50,000 cells/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2017-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (51):
- United States (8):
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Fort Worth, Texas
- Argentina (4):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
- Canada (5):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- Chile (2):
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- France (5):
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
- Germany (7):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Dortmund
- Italy (3):
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Monza, Lombardy
- Mexico (5):
  - GSK Investigational Site, Fracc. Las Americas, Aguascalientes
  - GSK Investigational Site, León, Guanajuato
  - GSK Investigational Site, DF
  - GSK Investigational Site, Durango
  - GSK Investigational Site, Mexico City
- Poland (4):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- GSK Investigational Site, Bloemfontein, Free State, South Africa
- Spain (4):
  - GSK Investigational Site, Alcalá de Henares
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santiago de Compostela
- United Kingdom (3):
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, London
  - GSK Investigational Site, Tooting, London

REFERENCES:
- [Derived] Morales-Ramirez J, Bogner JR, Molina JM, Lombaard J, Dicker IB, Stock DA, DeGrosky M, Gartland M, Pene Dumitrescu T, Min S, Llamoso C, Joshi SR, Lataillade M. Safety, efficacy, and dose response of the maturation inhibitor GSK3532795 (formerly known as BMS-955176) plus tenofovir/emtricitabine once daily in treatment-naive HIV-1-infected adults: Week 24 primary analysis from a randomized Phase IIb trial. PLoS One. 2018 Oct 23;13(10):e0205368. doi: 10.1371/journal.pone.0205368. eCollection 2018. PMID 30352054
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was originally designed for 96 weeks of treatment in treatment naïve human immunodeficiency virus-1 (HIV-1) infected adults; however, it was terminated early due to gastrointestinal intolerability and treatment emergent resistance. The study was conducted at 58 centers in 12 countries.
Pre-assignment Details: A total of 305 participants were screened, of which 210 were randomized to 1 of 4 treatment arms. Of 210 participants, only 206 received study treatment. Four participants were randomized but not treated as: 2 participants were randomized in error, 1 participant was lost to follow-up and 1 participant withdrew consent.
Groups:
- BMS-955176/GSK3532795 60 mg + TDF/FTC: Participants took one pill once daily from each of the three blinded bottles provided to them, containing BMS-955176/GSK3532795 60 milligrams (mg) active dose, BMS-955176/GSK3532795 placebo matching 120 mg and open-label tenofovir/emtricitabine (TDF/FTC) 300/200 mg from Day 1 to Week 96. The doses were administered in the morning with a meal. Participants took one pill once daily from the bottle containing efavirenz (EFV) placebo matching 600 mg at bed time on an empty stomach, without food from Day 1 to Week 96.
- BMS-955176/GSK3532795 120 mg + TDF/FTC: Participants took one pill once daily from each of the three blinded bottles provided to them, containing BMS-955176/GSK3532795 120 mg active dose, BMS-955176/GSK3532795 placebo matching 60 mg and open-label TDF/FTC 300/200 mg from Day 1 to Week 96. The doses were administered in the morning with a meal. Participants took one pill once daily from the bottle containing EFV placebo matching 600 mg at bed time on an empty stomach, without food, from Day 1 to Week 96.
- BMS-955176/GSK3532795 180 mg + TDF/FTC: Participants took one pill once daily from each of the three blinded bottles provided to them, containing BMS-955176/GSK3532795 60 mg active dose, BMS-955176/GSK3532795 120 mg active dose and open-label TDF/FTC 300/200 mg from Day 1 to Week 96. The doses were administered in the morning with a meal. Participants took one pill once daily from the bottle containing EFV placebo matching 600 mg once daily at bed time on an empty stomach, without food from Day 1 to Week 96.
- EFV 600 mg + TDF/FTC: Participants took one pill once daily from each of the three blinded bottles provided to them, containing BMS-955176/GSK3532795 placebo matching 60 mg, BMS-955176/GSK3532795 placebo matching 120 mg and open-label TDF/FTC 300/200 mg from Day 1 to Week 96. The doses were administered in the morning with a meal. Participants took one pill containing EFV 600 mg active dose once daily at bed time on an empty stomach, without food from Day 1 to Week 96.
Period: Overall Study
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC
Started | 50 | 52 | 51 | 53
Completed | 0 | 0 | 0 | 0
Not Completed | 50 | 52 | 51 | 53
Not completed — Administrative reason by sponsor | 39 | 40 | 41 | 39
Not completed — Adverse Event | 1 | 3 | 5 | 10
Not completed — Lack of Efficacy | 4 | 4 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 1 | 1
Not completed — Poor/Non-compliance | 1 | 0 | 1 | 0
Not completed — Reached stopping criteria | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 1 | 3
Not completed — Other | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics is presented for Treated Subjects Population, also known as the modified intent-to-treat (mITT) Population which comprised of all participants who received at least one dose of BMS-955176 or EFV.
Groups:
- BMS-955176/GSK3532795 60 mg + TDF/FTC: Participants took one pill once daily from each of the three blinded bottles provided to them, containing BMS-955176/GSK3532795 60 milligrams (mg) active dose, BMS-955176/GSK3532795 placebo matching 120 mg and open-label TDF/FTC 300/200 mg from Day 1 to Week 96. The doses were administered in the morning with a meal. Participants took one pill once daily from the bottle containing efavirenz (EFV) placebo matching 600 mg at bed time on an empty stomach, without food from Day 1 to Week 96.
- Total: Total of all reporting groups
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC | Total
Number analyzed (Participants) | 50 | 52 | 51 | 53 | 206
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated Subjects Population, also known as the modified intent-to-treat (mITT) population, comprised of all subjects who received at least one dose of study treatment, was used to present baseline characteristics
  Years | 31.8 (8.26) | 34.7 (11.29) | 35.5 (11.34) | 32.9 (9.35) | 33.7 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 7 | 7 | 30
  Male | 42 | 44 | 44 | 46 | 176
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race customized: White | 39 | 38 | 41 | 40 | 158
  Race customized: Black or African American | 8 | 10 | 6 | 9 | 33
  Race customized: American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Race customized: Unknown | 3 | 4 | 3 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Plasma HIV-1 Ribonucleic Acid (RNA) <40 Copies Per Milliliter (c/mL) at Week 24 Using Food and Drug Administration (FDA) Snapshot Algorithm
Description: Blood samples were collected for quantitative analysis of plasma HIV-1 RNA. The antiviral efficacy was determined by the number of participants with plasma HIV 1 RNA <40 c/mL at Week 24 using the FDA snapshot algorithm. This used the last on-treatment plasma HIV-1 RNA measurement within an FDA-specified visit window (18 to 30 weeks) to determine response. Analysis was performed on mITT Population, which comprised of randomized participants who received at least 1 dose of BMS-955176/GSK3532795 or EFV.
Time Frame: Week 24
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC
Number analyzed (Participants) | 50 | 52 | 51 | 53
Participants | 38 | 43 | 42 | 41

2. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA < 40 c/mL at Weeks 48 and 96 Using FDA Snapshot Algorithm
Description: Blood samples were collected for quantitative analysis of plasma HIV-1 RNA. The antiviral efficacy was determined by the number of participants with plasma HIV 1 RNA <40 c/mL at Weeks 48 and 96 using the FDA snapshot algorithm. This used the last on-treatment plasma HIV-1 RNA measurement within an FDA-specified visit window to determine response. The analysis was performed using mITT Population (observed), which consisted of participants in the mITT Population excluding participants who had no HIV-1 RNA result data in the assessment visit windows due to discontinuation and who discontinued on or after the date of site notification of study termination by the sponsor (10 October 2016). The data was not collected for Week 96 analysis; as the study was terminated early. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles).
Time Frame: Weeks 48 and 96
Population: mITT Population (observed)
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC
Number analyzed (Participants) | 50 | 52 | 51 | 53
Participants
  Week 48; n=40, 42, 40, 43: number analyzed (Participants) | 40 | 42 | 40 | 43
  Week 48; n=40, 42, 40, 43 | 35 | 41 | 40 | 40
  Week 96; n=0, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA < 200 c/mL at Week 24 Using FDA Snapshot Algorithm
Description: Blood samples were collected for quantitative analysis of plasma HIV-1 RNA. The antiviral efficacy was determined by the number of participants with plasma HIV-1 RNA <200 c/mL at Week 24 using the FDA snapshot algorithm. This used the last on-treatment plasma HIV-1 RNA measurement within an FDA-specified visit window to determine response.
Time Frame: Week 24
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC
Number analyzed (Participants) | 50 | 52 | 51 | 53
Participants | 40 | 44 | 43 | 44

4. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA < 200 c/mL at Weeks 48 and 96
Description: Blood samples were collected for quantitative analysis of plasma HIV-1 RNA. The antiviral efficacy was determined by the number of participants with plasma HIV-1 RNA <200 c/mL at Weeks 48 and 96 using the FDA snapshot algorithm. This used the last on-treatment plasma HIV-1 RNA measurement within an FDA-specified visit window to determine response. The analysis was performed using mITT Population (observed), which consisted of participants in the mITT Population excluding participants who had no HIV-1 RNA result data in the assessment visit windows due to discontinuation and who discontinued on or after the date of site notification of study termination by the sponsor (10 October 2016). The data was not collected for Week 96 analysis; as the study was terminated early. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles).
Time Frame: Weeks 48 and 96
Population: mITT Population (observed)
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC
Number analyzed (Participants) | 50 | 52 | 51 | 53
Participants
  Week 48; n=40, 42, 40, 43: number analyzed (Participants) | 40 | 42 | 40 | 43
  Week 48; n=40, 42, 40, 43 | 38 | 42 | 40 | 43
  Week 96; n=0, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Newly Emergent Genotypic Resistance Using All On-treatment Isolates
Description: The emergence of genotypic resistance among samples selected for drug resistance testing were assessed by searching for all reverse transcriptase substitutions and protease inhibitor substitutions listed in the International Acquired Immunodeficiency Syndrome (AIDS) Society-United States of America (IAS-USA) list of HIV-1 drug resistance mutations. The outcome was originally designed to be assessed up to 96 weeks of treatment, but it was analyzed up to Week 24 as the study was terminated early. The emergence of genotypic resistance is presented for participants in the mITT Population who had Baseline and on-treatment genotypic resistance testing and who had successful sequencing.
Time Frame: Week 24
Population: mITT Population. Only participants with Baseline and on-treatment genotypic resistance testing and who had successful sequencing were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC
Number analyzed (Participants) | 5 | 5 | 2 | 1
Participants
  Protease inhibitor substitution | 1 | 0 | 0 | 0
  Reverse transcriptase substitution | 3 | 5 | 2 | 0

6. Secondary Outcome: Number of Participants With Newly Emergent Phenotypic Resistance Using All On-treatment Isolates
Description: Phenotypic resistance to a drug is defined as a fold change (i.e., ratio of the 50% inhibitory concentration (IC50) of the clinical isolate to the IC50 of the reference strain) which is greater than the cut-off for reduced susceptibility. Emergent phenotypic resistance to BMS-955176/GSK3532795 was defined as a Baseline fold change IC50<= 3 and an on-treatment fold change IC50>3. The number of participants with newly emergent phenotypic resistance is presented for participants in the mITT Population who had Baseline and on-treatment phenotypic resistance testing. The outcome was originally designed to be assessed up to 96 weeks of treatment, but it was analyzed up to Week 24 as the study was terminated early.
Time Frame: Week 24
Population: mITT Population. Only participants who had Baseline and on-treatment phenotypic resistance testing were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC
Number analyzed (Participants) | 3 | 3 | 0 | 1
Participants | 1 | 0 |  | 0

7. Secondary Outcome: Change From Baseline in Logarithm to the Base 10 (log10) HIV-1 RNA Over Time
Description: Blood samples were collected for analysis of HIV-1 RNA. Values obtained at Day 1 were considered as Baseline value. Change from Baseline was calculated as value at indicated time point minus Baseline value. Change from Baseline in plasma HIV-1 RNA (log10) is summarized over time for the mITT Population using observed values, which excluded participants without HIV-1 RNA result data in the assessment visit windows due to discontinuation and who discontinued on or after the date of site notification of study termination by the sponsor (10 October 2016). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates standard deviation could not be calculated as only one participant was analyzed at the specified time point.
Time Frame: Baseline (Day 1) and Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72 and 84
Population: mITT Population (observed)
Measure: Mean (Standard Deviation); unit: Log 10 c/mL
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC
Number analyzed (Participants) | 50 | 52 | 51 | 53
Log 10 c/mL
  Week 2, n=8, 6, 10, 8: number analyzed (Participants) | 8 | 6 | 10 | 8
  Week 2, n=8, 6, 10, 8 | -1.927 (0.3726) | -1.930 (0.4785) | -2.006 (0.3783) | -2.003 (0.3662)
  Week 4, n=50, 51, 51, 50: number analyzed (Participants) | 50 | 51 | 51 | 50
  Week 4, n=50, 51, 51, 50 | -2.083 (0.5870) | -2.082 (0.5480) | -2.142 (0.5092) | -2.305 (0.4554)
  Week 8, n=49, 51, 49, 48: number analyzed (Participants) | 49 | 51 | 49 | 48
  Week 8, n=49, 51, 49, 48 | -2.308 (0.6989) | -2.262 (0.7152) | -2.334 (0.6046) | -2.516 (0.6408)
  Week 12, n=49, 50, 47, 47: number analyzed (Participants) | 49 | 50 | 47 | 47
  Week 12, n=49, 50, 47, 47 | -2.372 (0.8215) | -2.351 (0.7622) | -2.441 (0.6372) | -2.730 (0.6254)
  Week 16, n=47, 50, 46, 46: number analyzed (Participants) | 47 | 50 | 46 | 46
  Week 16, n=47, 50, 46, 46 | -2.502 (0.8650) | -2.432 (0.7991) | -2.513 (0.6429) | -2.862 (0.6903)
  Week 24, n=46, 47, 45, 44: number analyzed (Participants) | 46 | 47 | 45 | 44
  Week 24, n=46, 47, 45, 44 | -2.506 (0.8094) | -2.557 (0.7956) | -2.505 (0.7284) | -2.919 (0.7584)
  Week 32, n=44, 42, 42, 44: number analyzed (Participants) | 44 | 42 | 42 | 44
  Week 32, n=44, 42, 42, 44 | -2.497 (0.8045) | -2.642 (0.7408) | -2.528 (0.7392) | -2.920 (0.7488)
  Week 40, n=40, 42, 41, 43: number analyzed (Participants) | 40 | 42 | 41 | 43
  Week 40, n=40, 42, 41, 43 | -2.605 (0.7096) | -2.640 (0.7391) | -2.581 (0.6803) | -2.949 (0.7665)
  Week 48, n=40, 42, 40, 43: number analyzed (Participants) | 40 | 42 | 40 | 43
  Week 48, n=40, 42, 40, 43 | -2.650 (0.6824) | -2.649 (0.7388) | -2.557 (0.6711) | -2.935 (0.7415)
  Week 60; n=22, 24, 19, 20: number analyzed (Participants) | 22 | 24 | 19 | 20
  Week 60; n=22, 24, 19, 20 | -2.705 (0.6379) | -2.810 (0.5765) | -2.703 (0.7455) | -2.906 (0.5646)
  Week 72; n=5, 5, 5, 6: number analyzed (Participants) | 5 | 5 | 5 | 6
  Week 72; n=5, 5, 5, 6 | -2.586 (0.4682) | -2.733 (0.6809) | -2.725 (0.5025) | -2.780 (0.6598)
  Week 84; n= 2, 1, 2, 2: number analyzed (Participants) | 2 | 1 | 2 | 2
  Week 84; n= 2, 1, 2, 2 | -0.993 (3.4142) | -3.032 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -3.155 (0.1218) | -3.257 (0.5700)

8. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD)4+ Thymus (T)-Cell Counts Over Time
Description: CD4+ T-cell counts was assessed using flow cytometry. Values obtained at Day 1 were considered as Baseline value. Change from Baseline was calculated as value at indicated time point minus Baseline value. Change from Baseline in CD4+T- cell counts is summarized over time for the mITT Population using observed values, which excluded participants without HIV-1 RNA result data in the assessment visit windows due to discontinuation and who discontinued on or after the date of site notification of study termination by the sponsor (10 October 2016). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates standard deviation could not be calculated as only one participant was analyzed at the specified time point.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 60, 72 and 84
Population: mITT Population (observed)
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC
Number analyzed (Participants) | 50 | 52 | 51 | 53
Cells per microliter
  Week 4, n=50, 51, 50, 50: number analyzed (Participants) | 50 | 51 | 50 | 50
  Week 4, n=50, 51, 50, 50 | 41.6 (148.92) | 72.9 (167.53) | 52.9 (149.54) | 64.7 (145.51)
  Week 8, n=48, 49, 49, 47: number analyzed (Participants) | 48 | 49 | 49 | 47
  Week 8, n=48, 49, 49, 47 | 59.1 (219.64) | 81.8 (126.79) | 88.4 (177.68) | 117.4 (230.74)
  Week 12, n=49, 49, 47, 47: number analyzed (Participants) | 49 | 49 | 47 | 47
  Week 12, n=49, 49, 47, 47 | 110.4 (170.87) | 120.0 (178.04) | 129.7 (175.73) | 142.5 (118.39)
  Week 16, n=46, 50, 46, 46: number analyzed (Participants) | 46 | 50 | 46 | 46
  Week 16, n=46, 50, 46, 46 | 90.8 (200.76) | 99.7 (171.16) | 128.0 (212.09) | 140.5 (179.70)
  Week 24, n=46, 46, 44, 44: number analyzed (Participants) | 46 | 46 | 44 | 44
  Week 24, n=46, 46, 44, 44 | 94.3 (175.00) | 81.2 (195.39) | 92.5 (144.04) | 134.7 (151.70)
  Week 32, n=44, 42, 42, 44: number analyzed (Participants) | 44 | 42 | 42 | 44
  Week 32, n=44, 42, 42, 44 | 131.5 (207.69) | 103.5 (172.15) | 99.7 (171.95) | 175.6 (152.48)
  Week 40, n=41, 42, 41, 43: number analyzed (Participants) | 41 | 42 | 41 | 43
  Week 40, n=41, 42, 41, 43 | 175.9 (235.99) | 194.4 (235.14) | 167.3 (215.23) | 222.5 (191.99)
  Week 48, n=40, 41, 39, 43: number analyzed (Participants) | 40 | 41 | 39 | 43
  Week 48, n=40, 41, 39, 43 | 158.3 (228.90) | 152.0 (204.56) | 161.4 (221.65) | 232.4 (207.71)
  Week 60; n=22, 23, 19, 20: number analyzed (Participants) | 22 | 23 | 19 | 20
  Week 60; n=22, 23, 19, 20 | 168.4 (148.63) | 156.5 (301.91) | 198.3 (137.51) | 204.7 (154.86)
  Week 72; n=5, 5, 5, 7: number analyzed (Participants) | 5 | 5 | 5 | 7
  Week 72; n=5, 5, 5, 7 | 176.2 (98.50) | 336.8 (329.32) | 240.4 (240.48) | 209.7 (97.79)
  Week 84; n=2, 1, 2, 2: number analyzed (Participants) | 2 | 1 | 2 | 2
  Week 84; n=2, 1, 2, 2 | -4.0 (173.95) | 203.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 97.0 (285.67) | 165.5 (70.00)

9. Secondary Outcome: Change From Baseline in the Percentage of CD4+ T-cells Over Time
Description: CD4+ T-cell counts overall was assessed using flow cytometry. Values obtained at Day 1 were considered as Baseline value. Change from Baseline was calculated as value at indicated time point minus Baseline value. Change from Baseline in percentage of CD4+T- cell counts is summarized over time for the mITT Population using observed values, which excluded participants without HIV-1 RNA result data in the assessment visit windows due to discontinuation and who discontinued on or after the date of site notification of study termination by the sponsor (10 October 2016). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates standard deviation could not be calculated as only one participant was analyzed at the specified time point.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 60, 72 and 84
Population: mITT Population (observed)
Measure: Mean (Standard Deviation); unit: Percentage of CD4+T- cells
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC
Number analyzed (Participants) | 50 | 52 | 51 | 53
Percentage of CD4+T- cells
  Week 4, n=50, 51, 50, 50: number analyzed (Participants) | 50 | 51 | 50 | 50
  Week 4, n=50, 51, 50, 50 | 4.56 (3.195) | 3.43 (3.982) | 3.93 (3.210) | 3.87 (4.284)
  Week 8, n=48, 49, 49, 47: number analyzed (Participants) | 48 | 49 | 49 | 47
  Week 8, n=48, 49, 49, 47 | 5.02 (4.650) | 4.15 (4.047) | 5.15 (3.943) | 5.09 (4.257)
  Week 12, n=49, 49, 47, 47: number analyzed (Participants) | 49 | 49 | 47 | 47
  Week 12, n=49, 49, 47, 47 | 5.47 (4.570) | 5.39 (4.577) | 6.22 (4.450) | 6.29 (4.557)
  Week 16, n=46, 50, 46, 46: number analyzed (Participants) | 46 | 50 | 46 | 46
  Week 16, n=46, 50, 46, 46 | 6.20 (6.163) | 5.65 (4.179) | 6.95 (4.019) | 6.87 (4.763)
  Week 24, n=46, 46, 44, 44: number analyzed (Participants) | 46 | 46 | 44 | 44
  Week 24, n=46, 46, 44, 44 | 7.68 (5.834) | 5.71 (4.542) | 6.96 (4.761) | 5.94 (5.730)
  Week 32, n=44, 42, 42, 44: number analyzed (Participants) | 44 | 42 | 42 | 44
  Week 32, n=44, 42, 42, 44 | 7.75 (6.559) | 7.36 (5.457) | 6.90 (6.498) | 8.37 (6.253)
  Week 40, n=41, 42, 41, 43: number analyzed (Participants) | 41 | 42 | 41 | 43
  Week 40, n=41, 42, 41, 43 | 7.90 (6.612) | 6.97 (8.253) | 7.94 (5.601) | 9.06 (5.538)
  Week 48, n=40, 41, 39, 43: number analyzed (Participants) | 40 | 41 | 39 | 43
  Week 48, n=40, 41, 39, 43 | 9.07 (6.311) | 7.62 (6.218) | 9.59 (4.828) | 10.16 (6.262)
  Week 60; n=22, 23, 19, 20: number analyzed (Participants) | 22 | 23 | 19 | 20
  Week 60; n=22, 23, 19, 20 | 9.41 (6.290) | 8.44 (7.788) | 11.36 (6.568) | 10.73 (7.098)
  Week 72; n=5, 5, 5, 7: number analyzed (Participants) | 5 | 5 | 5 | 7
  Week 72; n=5, 5, 5, 7 | 8.56 (3.436) | 9.92 (4.147) | 12.46 (9.557) | 9.67 (3.982)
  Week 84; n=2, 1, 2, 2: number analyzed (Participants) | 2 | 1 | 2 | 2
  Week 84; n=2, 1, 2, 2 | -0.75 (8.839) | 4.60 (NA) — Standard deviation could not be analyzed as only one participant was analyzed. | 19.50 (11.314) | 12.90 (4.950)

10. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events Leading to Discontinuation (AELD)
Description: Any untoward medical occurrence that at any dose: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention were categorized as SAE. Number of participants with SAEs and AELDs is summarized.
Time Frame: Up to Week 96
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC
Number analyzed (Participants) | 50 | 52 | 51 | 53
Participants
  SAEs | 3 | 5 | 2 | 5
  AELD | 1 | 4 | 5 | 10

11. Secondary Outcome: Number of Participants With at Least One Centers for Disease Control (CDC) Class C Events
Description: The occurrence of new AIDS defining events that is CDC class C events is presented.
Time Frame: Up to Week 96
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC
Number analyzed (Participants) | 50 | 52 | 51 | 53
Participants | 0 | 2 | 0 | 0

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax), Observed Pre-dose Plasma Concentration (C0) and Observed Plasma Concentration at the End of a Dosing Interval (Ctau) of BMS-955176/GSK3532795
Description: Serial blood samples were collected at indicated time points for intensive pharmacokinetic (PK) assessment. The PK assessments were performed on evaluable PK Population, a sub-population which included all treated participants who had adequate PK profiles.
Time Frame: Pre-dose (morning) and at 0.5, 1, 1.5, 2, 4, 4.5, 5, 6, 8, 12 (evening pre-dose) and 24 hours (morning pre-dose) at Week 2 (Days 12 to 16)
Population: Evaluable PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC
Number analyzed (Participants) | 8 | 6 | 10
Nanogram per milliliter
  Cmax | 1945.342 (16.0) | 3162.161 (28.8) | 4645.266 (16.2)
  C0 | 1065.102 (25.2) | 1800.952 (33.4) | 2728.671 (17.8)
  Ctau | 1100.138 (15.1) | 1656.578 (39.7) | 2705.751 (26.8)

13. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of BMS-955176/GSK3532795
Description: Serial blood samples were collected at indicated time points for intensive PK assessment.
Time Frame: Pre-dose (morning) and 0.5, 1, 1.5, 2, 4, 4.5, 5, 6, 8, 12 (evening pre-dose) and 24 hours (morning pre-dose) at Week 2 (Days 12 to 16)
Population: Evaluable PK Population
Measure: Median (Full Range); unit: Hour
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC
Number analyzed (Participants) | 8 | 6 | 10
Hour | 4.00 [1.6 to 8.2] | 4.29 [4.0 to 5.1] | 5.50 [1.0 to 12.0]

14. Secondary Outcome: Area Under the Concentration-time Curve in One Dosing Interval (AUC [Tau]) of BMS-955176/GSK3532795
Description: Serial blood samples were collected at indicated time points for intensive PK assessment.
Time Frame: as for outcome 12
Population: Evaluable PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/ milliliter
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC
Number analyzed (Participants) | 8 | 6 | 10
Hour*nanogram/ milliliter | 34226.751 (18.73) | 55251.956 (32.88) | 87128.359 (20.79)

ADVERSE EVENTS:
Time Frame: Non-serious adverse events and serious adverse events (SAEs) were collected from the start of study treatment until Week 96.
Description: Non-SAEs and SAEs were collected in the mITT Population, which comprised of all participants who received at least one dose of BMS-955176/GSK3532795 or EFV.
Arm/Group | BMS-955176/GSK3532795 60 mg + TDF/FTC | BMS-955176/GSK3532795 120 mg + TDF/FTC | BMS-955176/GSK3532795 180 mg + TDF/FTC | EFV 600 mg + TDF/FTC
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/52 | 0/51 | 0/53
Serious Adverse Events (participants affected / at risk) | 3/50 | 5/52 | 2/51 | 5/53
Other Adverse Events (participants affected / at risk) | 41/50 | 46/52 | 45/51 | 48/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMS-955176/GSK3532795 60 mg + TDF/FTC (N=50) | BMS-955176/GSK3532795 120 mg + TDF/FTC (N=52) | BMS-955176/GSK3532795 180 mg + TDF/FTC (N=51) | EFV 600 mg + TDF/FTC (N=53)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic intolerance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMS-955176/GSK3532795 60 mg + TDF/FTC (N=50) | BMS-955176/GSK3532795 120 mg + TDF/FTC (N=52) | BMS-955176/GSK3532795 180 mg + TDF/FTC (N=51) | EFV 600 mg + TDF/FTC (N=53)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 6 (8) | 10 (14) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 3 (5) | 4 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 20 (30) | 22 (33) | 31 (58) | 8 (9)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 5 (6) | 2 (2) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 6 (7) | 7 (8)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (6) | 3 (4) | 2 (2)
Fatigue (General disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 4 (4) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 4 (5) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 6 (6) | 1 (1) | 3 (4)
Nasopharyngitis (Infections and infestations) | 5 (8) | 4 (5) | 6 (8) | 4 (4)
Pharyngitis (Infections and infestations) | 6 (7) | 3 (4) | 2 (4) | 3 (4)
Sinusitis (Infections and infestations) | 4 (5) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (7) | 8 (11) | 6 (8) | 1 (2)
Urethritis (Infections and infestations) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 21 (27)
Headache (Nervous system disorders) | 1 (1) | 6 (8) | 7 (8) | 6 (8)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 4 (5) | 1 (1) | 6 (6)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 1 (3) | 1 (1) | 7 (9) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 3 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.